CLINICAL TRIAL: NCT00624923
Title: Targeting Inflammation Using Salsalate in CardioVascular Disease (TINSAL-CVD)
Brief Title: Targeting Inflammation Using Salsalate in CardioVascular Disease
Acronym: TINSAL-CVD
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Joslin Diabetes Center (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other); Tufts Medical Center (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CHS 06-13; P50HL083813 (NIH); CCI: 2006-P-00175 (Other: Beth Israel Deaconess Medical Center, Boston, MA, USA); CHS: 06-13 (Other: Joslin Diabetes Center, Boston, MA, USA)
Record Dates: First submitted 2008-02-19; First posted 2008-02-28 (Estimated); Results first posted 2017-12-12 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-04

CONDITIONS: Coronary Artery Disease; Overweight
Keywords: Coronary Artery Disease; Inflammation; Overweight; Metabolic Syndrome; Salsalate
MeSH Terms: conditions — Coronary Artery Disease; Overweight; Inflammation; Metabolic Syndrome | interventions — salicylsalicylic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1- Active Pharmacologic (Experimental): Salsalate
  Interventions: Drug: Salsalate
- 2- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Salsalate — Salsalate, 500 mg, seven tablets daily by mouth, divided into two doses, for 30 months
  Other Names: Disalcid
  Arms: 1- Active Pharmacologic
Drug: Placebo — Placebo matched to Salsalate, seven tablets daily by mouth, divided into two doses, for 30 months
  Other Names: Placebo to Salsalate
  Arms: 2- Placebo

SUMMARY:
The hypothesis is that western lifestyle, with sedentary behaviors and caloric excess promote a chronic, subacute inflammatory state that participates in the development and progression of atherosclerosis. We will evaluate the effects of targeting inflammation using the anti-inflammatory drug salsalate, compared to placebo, on coronary artery plaque volume assessed by multi-detector computed tomographic angiography (MDCTA). The TINSAL-CVD study is a randomized, double-masked, placebo-controlled, 2 arm, clinical trial.

The purpose of the study is to compare the effect of salsalate or placebo on sub-acute inflammation and coronary plaque, in people with cardiovascular disease. Participants are randomized to active intervention (salsalate) or placebo interventions for a period of 30 months. The primary endpoint is change in plaque volume in the coronary arteries assessed by MDCTA from baseline to 30 months.

DETAILED DESCRIPTION:
OBJECTIVE:

To determine whether targeting inflammation using salsalate compared with placebo reduces progression of noncalcified coronary artery plaque.

DESIGN, SETTING, AND PARTICIPANTS:

In the Targeting Inflammation Using Salsalate in Cardiovascular Disease (TINSAL-CVD) trial participants were randomly assigned to 30 months of salsalate or placebo in addition to standard, guideline-based therapies. Randomization was computerized and centrally allocated, with patients, health care professionals, and researchers masked to treatment assignment. Participants were overweight and obese statin-using patients with established, stable coronary heart disease.

INTERVENTIONS:

Salsalate (3.5 g/d) or placebo orally over 30 months.

MAIN OUTCOMES AND MEASURES:

The primary outcome was progression of noncalcified coronary artery plaque assessed by multidetector computed tomographic angiography. Secondary outcomes were other measures of safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

Eligibility will be based upon the presence of established coronary artery disease including

* previous myocardial infarction (≥6 months ago), or
* previous coronary bypass surgery (> 12 months ago), or
* stable angina, or
* significant non-calcified plaque in at least one coronary artery, or
* abnormal exercise tolerance test or
* an area of reversible ischemia on nuclear imaging study or pharmacologic stress, with subsequent revascularization, or angioplasty, or
* abnormal exercise treadmill stress test with or without nuclear imaging or echocardiography with the following exclusions:

Exclusions based on nuclear imaging:

1. Transient cavity dilation
2. More than one vascular territory involved with reversible defect (multiple defects)
3. Reversible defects involving the anterior wall, septum or apex (LAD territory)

Exclusions based on echocardiography imaging:

1. More than one vascular territory involved with inducible wall motion abnormalities (multiple defects)
2. Inducible wall motion abnormalities involving the anterior wall, septum or apex (LAD territory)

Subjects should be at list 6 months after a myocardial infarction and/or revascularization procedure to be eligible.

In addition, subjects must be:

1. aged 21- 75 years inclusive,
2. BMI ≥ 27 kg/m2 and ≤ 35 kg/m2 if female and ≤ 40 kg/m2 if male (a BMI ≥24.5 for subjects from Asian origin)
3. on a stable dose of an HMG CoA reductase inhibitor (statin) for 1 month at screening or unable to tolerate a statin,
4. have normal renal function, (note estimated creatinine clearance calculated using Cockcroft-Gault (CG) equation ≥60 at screening [eCrCLCG (ml/min) = [(140 - age) x weight (kg)]/[SCr(mg/dl) x 72] x [0.85 if female],
5. have liver function (ALT, AST) < 3 times upper limits of normal),
6. normal thyroid function (on stable dose replacement therapy is acceptable),
7. if women are of child bearing potential they must have a pregnancy test prior to the CT angio and use contraception for the remainder of the study
8. patients with T2D must have a fasting glucose of ≤ 200 mg/dl at screening and cannot be treated with thiazolidinedione class agents or insulin or Extendin-4 (Byetta) therapy.

Subjects must be willing to have at least three visits at the Beth Israel-Deaconess Medical Center/Joslin Diabetes Center with a baseline and a 30-month follow-up series of imaging studies including CT angiography of the coronary arteries and imaging of the aorta, abdominal adiposity and liver, and interim visit at 1 year.

Exclusion Criteria:

1. Unstable angina (increase in frequency or severity of anginal episodes or development of chest pain at rest)
2. significant obstructive disease (≥ 70%) in left main coronary artery, ostial LAD or three-vessel disease by MDCTA
3. Significant heart failure (NYHA class III and IV)
4. Current atrial fibrillation or Wolf-Parkinson-White (WPW) syndrome
5. Allergy to beta-blocker in subjects with resting heart rate > 65 bpm
6. Systolic blood pressure > 160 mm Hg
7. Diastolic BP > 100 mm Hg
8. Persons with allergies to contrast material
9. History of asthma if unable to tolerate beta blocker
10. Allergy to iodinated contrast material or shellfish
11. Allergy to nitroglycerin
12. BMI > 35 kg/m2 if female and > 40 kg/m2 if male
13. Body weight > 350 lbs
14. Use of drugs for weight loss [e.g. Xenical (orlistat), Meridia (sibutramine), Acutrim (phenylpropanolamine) or similar over-the counter medications] within three months of screening
15. Surgery within 30 days of screening
16. History of acquired immune deficiency syndrome or human immunodeficiency virus (HIV)
17. Poor mental function or history of dementia/ Alzheimer's Disease or on medications used for treatment of dementia [e.g. Tacrine (Cognex), Rivastigmine (Exelon), Galantamine (Razadyne, Reminyl), Donepezil (Aricept), Memantine (Namenda)] or any other reason to expect patient difficulty in complying with the requirements of the study
18. Medicine for erectile dysfunction within 72 hours prior to MDCTA
19. History of significant chronic rheumatologic or other chronic inflammatory disease (including foot ulcers)
20. Prior hemorrhagic stroke
21. persons with known aspirin allergy
22. Use of continuous oral corticosteroid treatment (more than 2 weeks), or patients requiring corticosteroids within 3 months
23. Anti-diabetic medication including thiazolidinedione (pioglitazone or rosiglitazone), or insulin or Extendin-4 (Byetta)
24. History of peptic ulcer or gastritis within 5 years
25. Positive stool guaiac
26. Hemoglobin 2 standard deviations below normal
27. Low platelet count (2 standard deviations below normal)
28. Known bleeding disorder
29. Coumadin (warfarin compounds)
30. History of type 1 diabetes and/or history of ketoacidosis
31. Daily use of NSAIDS (including salsalate) for arthritis
32. History of malignancy, except subjects who have been disease-free for greater than 5 years, or whose only malignancy has been basal or squamous cell skin carcinoma
33. History of drug or alcohol abuse, or current weekly alcohol consumption >14 units/week (1 unit = 1 beer, 1 glass of wine, 1 mixed cocktail containing 1 ounce of alcohol)
34. Use of probenecid (Benemid, Probalan), sulfinpyrazone (Anturane) or other uricosuric agents
35. Chronic tinnitus.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Actual)
Dates: Start 2008-09 (Actual); Primary Completion 2015-01 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francine Welty, MD, Study Director — Beth Israel Deaconess Medical Center; Allison B. Goldfine, MD, Principal Investigator — Joslin Diabetes Center; Ernest Schaefer, MD, Principal Investigator — Tufts Medical Center; Melvin Clouse, MD, Principal Investigator — Beth Israel Deaconess Medical Center; Steven E. Shoelson, MD, PhD, Principal Investigator — Joslin Diabetes Center
Locations (5):
- United States (5):
  - Seacoast Cardiology, York Village, Maine
  - Joslin Diabetes Center, Boston, Massachusetts
  - Heart Center of Metrowest, Framingham, Massachusetts
  - South Shore Internal Medicine, Milton, Massachusetts
  - Newton-Wellesley Cardiology, Newton, Massachusetts

REFERENCES:
- [Background] Shoelson SE, Lee J, Goldfine AB. Inflammation and insulin resistance. J Clin Invest. 2006 Jul;116(7):1793-801. doi: 10.1172/JCI29069. PMID 16823477
- [Background] Fleischman A, Shoelson SE, Bernier R, Goldfine AB. Salsalate improves glycemia and inflammatory parameters in obese young adults. Diabetes Care. 2008 Feb;31(2):289-94. doi: 10.2337/dc07-1338. Epub 2007 Oct 24. PMID 17959861
- [Background] Goldfine AB, Silver R, Aldhahi W, Cai D, Tatro E, Lee J, Shoelson SE. Use of salsalate to target inflammation in the treatment of insulin resistance and type 2 diabetes. Clin Transl Sci. 2008 May;1(1):36-43. doi: 10.1111/j.1752-8062.2008.00026.x. PMID 19337387
- [Background] Goldfine AB, Fonseca V, Jablonski KA, Pyle L, Staten MA, Shoelson SE; TINSAL-T2D (Targeting Inflammation Using Salsalate in Type 2 Diabetes) Study Team. The effects of salsalate on glycemic control in patients with type 2 diabetes: a randomized trial. Ann Intern Med. 2010 Mar 16;152(6):346-57. doi: 10.7326/0003-4819-152-6-201003160-00004. PMID 20231565
- [Background] Goldfine AB, Fonseca V, Jablonski KA, Chen YD, Tipton L, Staten MA, Shoelson SE; Targeting Inflammation Using Salsalate in Type 2 Diabetes Study Team. Salicylate (salsalate) in patients with type 2 diabetes: a randomized trial. Ann Intern Med. 2013 Jul 2;159(1):1-12. doi: 10.7326/0003-4819-159-1-201307020-00003. PMID 23817699
- [Background] Goldfine AB, Conlin PR, Halperin F, Koska J, Permana P, Schwenke D, Shoelson SE, Reaven PD. A randomised trial of salsalate for insulin resistance and cardiovascular risk factors in persons with abnormal glucose tolerance. Diabetologia. 2013 Apr;56(4):714-23. doi: 10.1007/s00125-012-2819-3. Epub 2013 Jan 31. PMID 23370525
- [Background] Avadhani R, Fowler K, Barbato C, Thomas S, Wong W, Paul C, Aksakal M, Hauser TH, Weinger K, Goldfine AB. Glycemia and cognitive function in metabolic syndrome and coronary heart disease. Am J Med. 2015 Jan;128(1):46-55. doi: 10.1016/j.amjmed.2014.08.025. Epub 2014 Sep 16. PMID 25220612
- [Background] Goldfine AB, Shoelson SE. Therapeutic approaches targeting inflammation for diabetes and associated cardiovascular risk. J Clin Invest. 2017 Jan 3;127(1):83-93. doi: 10.1172/JCI88884. Epub 2017 Jan 3. PMID 28045401
- [Background] Ridker PM. Informative Neutral Studies Matter-Why the Targeting Inflammation With Salsalate in Cardiovascular Disease (TINSAL-CVD) Trial Deserves Our Attention. JAMA Cardiol. 2016 Jul 1;1(4):423-4. doi: 10.1001/jamacardio.2016.0604. No abstract available. PMID 27438318
- [Result] Hauser TH, Salastekar N, Schaefer EJ, Desai T, Goldfine HL, Fowler KM, Weber GM, Welty F, Clouse M, Shoelson SE, Goldfine AB; Targeting Inflammation Using Salsalate in Cardiovascular Disease (TINSAL-CVD) Study Team. Effect of Targeting Inflammation With Salsalate: The TINSAL-CVD Randomized Clinical Trial on Progression of Coronary Plaque in Overweight and Obese Patients Using Statins. JAMA Cardiol. 2016 Jul 1;1(4):413-23. doi: 10.1001/jamacardio.2016.0605. PMID 27438317
- [Derived] Day EA, Ford RJ, Smith BK, Houde VP, Stypa S, Rehal S, Lhotak S, Kemp BE, Trigatti BL, Werstuck GH, Austin RC, Fullerton MD, Steinberg GR. Salsalate reduces atherosclerosis through AMPKbeta1 in mice. Mol Metab. 2021 Nov;53:101321. doi: 10.1016/j.molmet.2021.101321. Epub 2021 Aug 21. PMID 34425254
- See also: This site provides information on a related clinical trial to target inflammation using salsalate to lower blood glucose in patients with type 2 diabetes mellitus. — http://tinsalt2d.org
- See also: Home page for Joslin Diabetes Center, Boston, MA. — http://joslin.org

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 340 subjects signed consent and were screened for eligibility.
Groups:
- 2- Placebo: Placebo
  Placebo: Salsalate Placebo, seven tablets daily by mouth, divided into two doses, for 30 months
Period: Overall Study
Arm/Group | 1- Active Pharmacologic | 2- Placebo
Started | 127 | 124
Completed | 89 | 101
Not Completed | 38 | 23

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1- Active Pharmacologic | 2- Placebo | Total
Number analyzed (Participants) | 127 | 124 | 251
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.5 (6.8) | 60.1 (7.2) | 60.8 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 15
  Male | 118 | 118 | 236
Region of Enrollment [Number; unit: participants]
  United States | 127 | 124 | 251
Statin use [Number; unit: participants] | 126 | 122 | 248

OUTCOME MEASURES:

1. Primary Outcome: Change in Non-calcified Plaque Volume in the Coronary Arteries Assessed by MDCTA From Baseline to 30 Months
Time Frame: Baseline to 30 months
Population: Intention to Treat
Measure: Mean (95% Confidence Interval); unit: mm^3
Groups:
- 2-Placebo: Placebo
  Placebo: Salsalate Placebo, seven tablets daily by mouth, divided into two doses, for 30 months
Arm/Group | 1- Active Pharmacologic | 2-Placebo
Number analyzed (Participants) | 84 | 89
mm^3 | 0 [-8 to 7] | 0 [-7 to 7]

2. Secondary Outcome: Change in Cholesterol
Description: secondary
Time Frame: Baseline to 30 mo
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | 1- Active Pharmacologic | 2- Placebo
Number analyzed (Participants) | 127 | 124
mg/dL | 5.1 [1.2 to 9.0] | 2.0 [-1.7 to 5.6]

3. Secondary Outcome: Change in Inflammation Marker: CRP
Description: Secondary outcome of change in inflammation marker CRP
Time Frame: baseline to 30 mo
Measure: Mean (95% Confidence Interval); unit: mg/L
Arm/Group | 1- Active Pharmacologic | 2- Placebo
Number analyzed (Participants) | 127 | 124
mg/L | -0.1 [-0.4 to 0.2] | -0.1 [-0.4 to 0.1]

4. Secondary Outcome: Change in Inflammation in the Liver Associated With Nonalcoholic Steatohepatitis (NASH), ALT
Description: Secondary outcome, change in liver inflammation associated with NASH: ALT
Time Frame: baseline to 30 mo
Measure: Mean (95% Confidence Interval); unit: U/L
Arm/Group | 1- Active Pharmacologic | 2- Placebo
Number analyzed (Participants) | 127 | 124
U/L | -1.1 [-2.1 to -0.1] | -0.6 [-1.6 to 0.4]

ADVERSE EVENTS:
Description: Standard FDA definitions of AE/SAE used.
Arm/Group | 1- Active Pharmacologic | 2- Placebo
Serious Adverse Events (participants affected / at risk) | 33/127 | 32/124
Other Adverse Events (participants affected / at risk) | 127/127 | 112/124
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 1- Active Pharmacologic (N=127) | 2- Placebo (N=124)
Cardiac (Cardiac disorders) | 13 | 19
Vascular (Blood and lymphatic system disorders) | 3 | 2
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 5 | 4
Gastrointestinal (Gastrointestinal disorders) | 4 | 6
Renal (Renal and urinary disorders) | 5 | 0
Hepatobiliary (Hepatobiliary disorders) | 1 | 1
Infectious (Infections and infestations) | 3 | 1
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Dermatologic (Skin and subcutaneous tissue disorders) | 1 | 0
General (General disorders) | 3 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 1- Active Pharmacologic (N=127) | 2- Placebo (N=124)
Ear and Labyrinth (Ear and labyrinth disorders) | 35 | 13
General (General disorders) | 17 | 13
Gastrointestinal (Gastrointestinal disorders) | 15 | 9
Respiratory (Respiratory, thoracic and mediastinal disorders) | 64 | 54
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 21 | 15
Mouth sores (Gastrointestinal disorders) | 13 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No